CLINICAL TRIAL: NCT06137430
Title: Effect of Sodium Glucose Cotransporter 2 Inhibitiors on Left Ventricular Remodeling Among Diabetic and Non Diabetic Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Abd eltwab Abd elzaher, Ahmad Abd eltwab Abd elzaher, Assiut University
Other Study IDs: Effect of SGLT2 inhibitiors
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: SGLT2 Inhibitiors Remodeling Effect; Chronic Heart Disease
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Diabetic patients with chronic heart failure
  Interventions: Drug: Sodium-glucose cotransporter 2 inhibitor
- Non_diabetic patients with chronic heart failure
  Interventions: Drug: Sodium-glucose cotransporter 2 inhibitor

INTERVENTIONS:
Drug: Sodium-glucose cotransporter 2 inhibitor — Sodium glucose cotransporter 2 inhibitiors

SUMMARY:
To evaluate the efficacy of SGLT2 inhibitors on left ventricular global longitudinal strain and diastology parameters among diabetic and non-diabetic patients with chronic heart failure

DETAILED DESCRIPTION:
Sodium-glucose cotransporter 2 inhibitors (SGLT2i) have an established place in the therapy of heart failure (HF), as they have been shown to significantly reduce all-cause mortality, cardiovascular mortality, and hospitalizations in HFrEF patients, regardless of the presence of diabetes mellitus.

The growing evidence of the effect of SGLT2i on cardiac remodeling through cellular, molecular, vascular, interstitial, and electrical effects justifies its role as fundamental HF therapy.

SGLT2 inhibition in heart failure promotes reverse cardiac remodeling and is associated with better clinical outcomes.

Adverse myocardial remodeling affecting the left ventricle is a key factor in HF progression, and current well-established HF phenotypes are based on LVEF. However, other relevant players, such as the left atrium, have received less attention. Indeed, the left atrium plays a critical role in cardiac function, particularly in left ventricular (LV) filling during diastole. Additionally, atrial dysfunction can directly lead to pulmonary congestion. Left atrial (LA) remodeling occurs in HF irrespective of the degree of LV systolic dysfunction and can be observed in the presence of preserved or reduced LVEF. SGLT2 inhibition has been associated with reduced left ventricular (LV) and left atrial volumes in HF; however, its relationship with contemporary echocardiographic parameters of global LV systolic function, including global longitudinal strain and myocardial work, has not been thoroughly investigated.

Measuring the effect of SGLT2i therapy on left ventricular systolic function (LV) has previously been assessed by changes in heart size volume and ejection fraction.

In current clinical practice, the assessment of LV systolic function is still mainly based on the measurement of LV ejection fraction (LVEF), which remains the gold standard despite some notable limitations.

In the last decade, LV global longitudinal strain (GLS) has emerged as a more accurate predictor of poor outcomes, revealing subtle abnormalities and preclinical LV systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

- The study will enroll outpatients with HF on optimized medical therapy defined by the guidelines of the European Society of Cardiology (ESC) that were used when the study was initiated.

Age ranges from 18 to 75 years

Exclusion Criteria:

* age <18 and > 75 years. 2. If there is any contraindication in using SGLT2 inhibitors, patients that had symptomatic hypotension (systolic blood pressure < 95 mmHg, impaired renal function (eGFR <30ml/min/1.73m2 calculated by the CKD-EPI formula), Potassium serum levels > 5.2 mmol/L and Liver dysfunction (defined as hepatic parameters such as ALT, AST and/or ALP elevated ≥3 times above the upper 99th reference percentile.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: diabetic and non-diabetic with chronic heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular global longitudinal strain and diastology parameters, including (left atrial volume indexed) LAVI in chronic heart failure patients on SGLT2 inhibitors, comparing diabetic and non-diabetic patients | Baseline
  Effect of SGLT2 inhibitiors on left ventricular remodeling among diabetic and non diabetic patients with chronic heart failure